CLINICAL TRIAL: NCT00210249
Title: Development of an Evaluation Method of Elderly Condition in Patient Receiving Chemotherapy Treatment . Geriatric Oncology Protocol in Aquitaine Country.
Brief Title: Development of an Evaluation Method of Elderly Condition in Patient Receiving Chemotherapy Treatment
Acronym: PHRC2003
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: Sanofi-Synthelabo (Industry); Aventis Pharmaceuticals (Industry); Amgen (Industry); Chugai Pharmaceutical (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IB2002-26; PHRC OncoG (Other: Institut Bergonié)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2022-01-12 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Lymphoma; Digestive System Diseases; Ovarian Diseases; Pulmonary Disease; Prostatic Disease; Bladder Disease
Keywords: Cancer; elderly; geriatric evaluation; safety; chemotherapy
MeSH Terms: conditions — Lymphoma; Digestive System Diseases; Ovarian Diseases; Lung Diseases; Prostatic Diseases; Urinary Bladder Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Incidence of cancer in 75+ years old is 16,500 new cases per year, more than fifty percent of people with cancerThey are very few therapeutic trials dedicated. Oncologists hesitate to treat them because they are either afraid of inducing toxicity or of breaking down quality of life. Consequently, we decided to launch a protocol with both oncologists and geriatricians which principal aim is to find out if geriatric assessment data can help to better predict for chemotherapy toxicity, loss of autonomy and survival. We plan to accrue 360 patients diagnosed for cancer, including digestive, pulmonary, prostate, lymphoma, bladder, ovary cancer for whom first-line chemotherapy is planned. Patients are initially classified according to usual methods of medical oncology practice into three groups: patients who can receive standard treatment, reduced standard treatment or treatment adapted to the frail condition. Around Aquitaine, , we organised seven teams composed of one geriatrician and one nurse. Two kind of teams were activated: one which cover ten treatment sites in Bordeaux area and six sedentary teams which worked half a day a week in designated hospitals . Geriatric evaluation included test of cognitive functions (MMS), nutritional status (MNA), co-morbidity (CIRS-G), mobility (Get up and Go), activities (ADL;IADL), quality of life (QLQ-C30), depression (GDS-15) and Lachs-Balducci screening. Patients have four geriatric evaluations : before treatment, day 1 cycle 2, day 1 cycle 4, day 1 cycle 7 and/or end of chemotherapy. Since September 2002, 177 patients have been included, 112 have finished: 47.3% have received four evaluations, 16.1% died before the end of protocol, 14.3% stopped because they were in progression and changed their treatment, 11.6% met administrative problem that didn't allow all evaluations, 7.1% declined after inclusion and 3.6% finished their treatment before. The following results have been obtained: before treatment, 73% of these patients were at risk of undernutrition (MNA< 23.5), about 1/3 had one or more inability or a risk of falls (38% IADL<6, 29% get up and go>20seconds, 27% ADL>1, 34% PS<1), 28% of them had altered cognitive functions (MMS<24), 29% were depressive (GDS-15>6), 25% thought they had poor quality of life (QLQ-C30<4). Protocol will be closed in September 2005.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 70 years
* First line of chemotherapy
* Cancer previously mentioned

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients greater than 70 year of age (no upper age limit) who were scheduled to receive first-line chemotherapy for various types of cancer (ie, colon, pancreas, stomach, ovary, bladder, prostate, lung cancer, non-Hodgkin's lymphoma [NHL], or cancer of unknown primary origin), excluding breast cancer, were eligible for inclusion. Patients with known CNS metastases were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2002-09 (Actual); Primary Completion 2007-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre SOUBEYRAN, MD, PhD, Principal Investigator — Institut Bergonié
Locations (18):
- France (18):
  - Centre de radiothérapie d'Agen, Agen
  - Centre Hospitalier Universitaire d'Agen, Agen
  - Clinique Esquirol Saint Hilaire, Agen
  - Centre Hospitalier Universitaire de Bayonne, Bayonne
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Clinique Saint Etienne du Pays Basque, Bayonne
  - Clinique Tivoli, Bordeaux
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Institut Bergonié - Centre Régional de Luttre Contre le Cancer de Bordeaux et du Sud Ouest, Bordeaux
  - Centre Hospitalier Universitaire de Dax, Dax
  - Hopital Sub-Urbain du Bouscat, Le Bouscat
  - Hôpital Robert Boulin, Libourne
  - Centre Hospitalier Universitaire de Mont de Marsan, Mont-de-Marsan
  - Centre Hospitalier Universitaire de Pau, Pau
  - Centre Hospitalier Universitaire de Perigueux, Périgueux
  - Clinique Francheville, Périgueux
  - Maison de Santé Protestante Bagatelle, Talence
  - Centre Hospitalier Universitaire de Villeneuve sur Lot, Villeneuve-sur-Lot

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Soubeyran P, Fonck M, Blanc-Bisson C, Blanc JF, Ceccaldi J, Mertens C, Imbert Y, Cany L, Vogt L, Dauba J, Andriamampionona F, Houede N, Floquet A, Chomy F, Brouste V, Ravaud A, Bellera C, Rainfray M. Predictors of early death risk in older patients treated with first-line chemotherapy for cancer. J Clin Oncol. 2012 May 20;30(15):1829-34. doi: 10.1200/JCO.2011.35.7442. Epub 2012 Apr 16. PMID 22508806
- [Derived] Hoppe S, Rainfray M, Fonck M, Hoppenreys L, Blanc JF, Ceccaldi J, Mertens C, Blanc-Bisson C, Imbert Y, Cany L, Vogt L, Dauba J, Houede N, Bellera CA, Floquet A, Fabry MN, Ravaud A, Chakiba C, Mathoulin-Pelissier S, Soubeyran P. Functional decline in older patients with cancer receiving first-line chemotherapy. J Clin Oncol. 2013 Nov 1;31(31):3877-82. doi: 10.1200/JCO.2012.47.7430. Epub 2013 Sep 23. PMID 24062399

RESULTS

PARTICIPANT FLOW:
Groups:
- Eligible Patients: Patients satisfying eligibility criteria
Period: Overall Study
Arm/Group | Eligible Patients
Started | 364
Completed | 348
Not Completed | 16
Not completed — Lost to Follow-up | 5
Not completed — Protocol Violation | 11

BASELINE CHARACTERISTICS:
Arm/Group | Eligible Patients
Number analyzed (Participants) | 364
Age, Continuous [Median (Full Range); unit: years] | 77.45 [70 to 99.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157
  Male | 207
Region of Enrollment [Number; unit: participants]
  France | 364

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant Deaths
Description: Number of participant deaths observed during the course of the study
Time Frame: 6 months after inclusion
Population: Eleven patients did not complete the geriatric evaluation, and an additional five patients were lost to follow-up before 6 months, which left 348 analyzed patients
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Patients
Number analyzed (Participants) | 348
Participants | 56

ADVERSE EVENTS:
Time Frame: Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Eligible Patients
All-Cause Mortality (participants affected / at risk) | 56/348
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No